CLINICAL TRIAL: NCT05321615
Title: A Prospective Study to Assess the Feasibility and Safety of a Wireless Palpator to Detect Occult Subpleural Lung Tumours in Humans During Minimally Invasive (VATS) Lung Resection.
Brief Title: Feasibility and Safety of a Wireless Palpator
Acronym: Palpator
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Richard Malthaner, Chair Chief Thoracic Surgery, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Palpator 2022-02-22
Record Dates: First submitted 2022-02-23; First posted 2022-04-11 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Lung Cancer; Thoracic Neoplasm
Keywords: Palpation; Tactile image sensor; Lung ultrasound; VATS procedures
MeSH Terms: conditions — Lung Neoplasms; Thoracic Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Other): All patients will undergo a standard VATS pleuroscopy to visually search for the nodule and its position. Sequential assessment using a grasper, the Palpator, the VATS ultrasound probe, and then finger palpation will be done to detect the nodule.
  Interventions: Device: Palpator; Device: Grasper; Device: Ultrasound; Other: Finger palpation

INTERVENTIONS:
Device: Palpator — Palpator for tumor localization
Device: Grasper — Atraumatic lung grasper
Device: Ultrasound — VATS ultrasound
Other: Finger palpation — Palpation of the lung/tumour using the surgeon's finger

SUMMARY:
Evaluation of the ability of the Palpator to detect hidden (occult) lung tumours that cannot be visualized or palpated using the traditional methods of visual inspection, grasper palpation, and VATS ultrasound.

DETAILED DESCRIPTION:
All procedures will be performed with the patient under general anesthesia with single lung ventilation through double-lumen endotracheal intubation. Three to four thoracoports, no larger than 12 mm, will be inserted in the intercostal spaces as needed. After VATS port placement, the pleural cavity will be insufflated with CO2 to a maximum pressure of 8 mm Hg to assist with lung deflation. A standard VATS pleuroscopy will be performed to visually search for the nodule and its position confirmed with sequential assessment using a grasper, the Palpator, the VATS ultrasound probe, and then finger palpation. This will ensure that all patients will have the opportunity to avoid a large thoracotomy if the lesion can't be identified by the Palpator. If the lesion can be detected either visually or by grasper palpation, this information will be recorded, but will be excluded from the analysis of Palpator feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Peripheral occult sub-pleural (>5 mm) solitary lung nodule < 50 mm on CT scan scheduled for surgical removal using a VATS approach

Exclusion Criteria:

* Semi-solid nodules (ground glass nodule).
* Pregnancy or potentially pregnant women.
* Mentally challenged.
* Inability to consent for the study.
* Patients less than 18 years old.
* Patients with pulmonary nodules easily located during VATS (> 50 mm, pleural puckering, invading chest wall)
* Patients who have chest anatomy precluding VATS resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Tumour detection | 1 day
  The palpator will be declared feasible of it can detect at least 80% of tumours (sensitivity) without the need for a thoracotomy.

SECONDARY OUTCOMES:
Prevention of thoracotomy | 1 day
  The number of patients undergoing conversion from VATS to open thoracotomy
Adverse events | 30 days
  Adverse events will be recorded.

IPD SHARING:
Plan to Share IPD: No
no plan